CLINICAL TRIAL: NCT04087954
Title: Evaluation the Impact of Self-Stigma Reduction Program on Psychosocial Outcomes Among People Diagnosed With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fakeeh College for Medical Sciences (Other)
Responsible Party: Principal Investigator, Abd Alhadi Hasan, Assistant professor, Fakeeh College for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5115
Record Dates: First submitted 2019-09-07; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Stigmatization
MeSH Terms: conditions — Stereotyping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention vs control (Experimental)
  Interventions: Behavioral: Stigma reduction program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Stigma reduction program — Participants in the intervention group received treatment as usual, supported with stigma reduction program booklets each fortnight for 26 weeks. The stigma reduction program includes three modules; psychoeducation, cognitive behavioural therapy and social skills training. The program aims to enhance patient understanding of Schizophrenia and foster communication skills which supposed to increase self-confidence and strengthen communication networking with society.
  Psychoeducation module purposes at introducing about the concepts of schizophrenia, providing patient with essential information about schizophrenia, including nature of disease, sign/symptoms, treatment strategies, side effects of medication. Social Skills Training (SST) module purposes at fostering communication skills among patient diagnosed with schizophrenia. This assists the participants to be re-integrated in the society and build a harmonious atmosphere in the community.
  Arms: Intervention vs control

SUMMARY:
Backgrounds: Research evidence suggests that people diagnosed with schizophrenia (PDwS) experience higher level of stigma compared with other forms of mental illness, and they are prone to internalize stereotype, which exacerbates severity of psychiatric symptoms, reduces their psychosocial treatment adherence. The purpose of the study to evaluate the effectiveness of stigma reduction program on the perceived stigma, psychiatric symptoms, compliance with psychosocial intervention and self-efficacy.

Methods: A randomized controlled trial was conducted from November 2017 to December 2018 with 278 PDwS. Participants aged 18 years or older with DSM-IV schizophrenia or schizoaffective disorder, from four outpatient mental health clinics in Jordan, were randomly assigned to receive 13 sessions of a booklet form of stigma reduction program (n = 140) (psycho-education, cognitive behavioural therapy and social skills training), and treatment as usual [TAU] (intervention, n = 140), or TAU (control, n = 138). Participants were assessed at baseline, immediately post-intervention (post-treatment1) and at six months follow-up. The primary outcome measure was change in stigma perception. Secondary outcomes were psychiatric symptoms, compliance with psychosocial interventions and self-efficacy.

ELIGIBILITY:
Eligibility Criteria

* Adults aged 18 or over diagnosed with schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) (American Psychiatric Association, 2013).
* All participants had to be able to read and write English or Arabic
* Willing and able to consent.

Exclusion criteria were:

- People diagnosed with schizophrenia who had a learning disability, with known organic mental disorder, substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
The primary outcome was stigma perception measured by the Internalised Stigma of Mental Illness Scale (ISMI) | November 2017-December 2018 (up to 11 months)
  The primary outcome was stigma perception measured by the Internalised Stigma of Mental Illness Scale (ISMI). This scale has 29 items measure service user experience of stigma. It is composed of 5 subscales: alienation (6 items), stereotype endorsement (7 items), discrimination experience (5 items), social withdrawal (6 items), and stigma resistance (5 items). Each item is rated on a four-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). The five stigma resistance subscale items are reverse-coded, and also serve as a validity check. The stigma resistance score is calculated by subtracting the actual value from five. Therefore, stigma resistance displays the same direction of correlation as the other four subscales. A high total score on the ISMI scale indicates more severe internalized stigmatization. The internal consistency is (α=0.90) and test-retest reliability (r=0.92) have been reported for the ISMI (Ritsher & Phelan, 2004).

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) | November 2017-December 2018 (up to 11 months)
  PANSS measures 30 clinical symptoms of schizophrenia; each symptom is scored from 1 indicating absence of psychopathology to 7 indicating severe psychopathology, with higher scores indicating poorer mental health status. Internal reliability and criterion-related validity are 0.77 (positive scale) and 0.77 (negative scale), and 0.52 with the Clinical Global Impression scale (CGI) (Kay, Fiszbein, & Opfer, 1987). The primary researcher (AH) attended training delivered by the PANSS Institute, USA, and trained the outcomes assessors. An inter-rater reliability checked prior to the study, between assessors was 0.75 and inter-rater reliability (intra-class correlation (ICC) was 0.79. This tool was administered in English by the primary researcher (AH) and research assistants.
The Psychosocial Treatment Compliance Scale (PTCS) | November 2017-December 2018 (up to 11 months)
  The Psychosocial Treatment Compliance Scale (PTCS) (Tsang et al., 2006) has 17 items rated from "(1) never" to "(5) always". The PTCS has the "participation" (12 items) and "attendance" (5 items) subscales. The scale has two main parts, participation which indicates the level of participants engagement and participation in the psychosocial interventions (e.g., "was willing to follow therapists' instructions"). However, attendance measures that participants commitment to scheduled appointments (e.g., "attended prescribed psychosocial treatment on time"). The scale has good psychometric properties (internal consistency: α=.87-.96; test-retest reliability: ICC=.86-.90) were demonstrated for the subscales (Tsang et al., 2006).
The Chinese General Self-efficacy Scale (CGSS) | November 2017-December 2018 (up to 11 months)
  The Chinese General Self-efficacy Scale (CGSS) developed by (Chiu & Tsang, 2004). This scale has a 10-item. Scoring system ranges from "(1) Not at all true" to "(4) Exactly true". Participants with higher score reflect better general self-efficacy. The CGSS demonstrated good internal consistency (α=0.92-0.93) and test-retest reliability (ICC=0.75-0.94) (Chiu & Tsang, 2004).

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasan AA, Alasmee N. Evaluation of the impact of a self-stigma reduction programme on psychosocial outcomes among people with schizophrenia spectrum disorder. J Ment Health. 2022 Feb;31(1):83-91. doi: 10.1080/09638237.2021.1922628. Epub 2021 Sep 14. PMID 34517747